CLINICAL TRIAL: NCT03186768
Title: Evaluation of Soap on a Rope Hall Pass Behavior Intervention: a School-randomized Controlled Trial
Brief Title: Soap on a Rope Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Syracuse University (Other)
Responsible Party: Principal Investigator, David Larsen, Assistant Professor, Syracuse University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SoapRopetrial
Record Dates: First submitted 2017-05-18; First posted 2017-06-14 (Actual); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Hand Disinfection

STUDY DESIGN:
Intervention Model Description: School-randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: School group (intervention or control) will be blinded for data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Intervention arm receives a training of trainers on the soap on a rope hall pass intervention.
  Interventions: Behavioral: Soap on a rope hall pass intervention
- Control arm (No Intervention): Control arm delays the training of trainers on the soap on a rope hall pass intervention until endline hand washing data has been collected.

INTERVENTIONS:
Behavioral: Soap on a rope hall pass intervention — School health and nutrition coordinators will be trained on how to make and utilize the soap on a rope hall pass to improve hand washing behavior in schools.
  Arms: Intervention arm

SUMMARY:
The soap on a rope behavioral trial is a school-randomized trial to determine if a disruptive cue (the soap on a rope hall pass) can influence hand washing behavior for students in Namwala District, Zambia.

ELIGIBILITY:
Inclusion Criteria:

* Students in study schools who use the latrine on the day of observation

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Change in hand washing behavior | Handwashing behavior will be monitored at three time points: baseline, 3 weeks following the intervention, and 8 weeks following the intervention.
  Students exiting the latrine will be monitored to determine if they wash their hands using soap and water.

CONTACTS AND LOCATIONS:
Overall Officials: David A Larsen, PhD, MPH, Principal Investigator — Syracuse University
Locations (1):
- Namwala District, Namwala, Zambia

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared upon reasonable request. Email Dr. David Larsen at dalarsen@syr.edu.